CLINICAL TRIAL: NCT03880136
Title: A Phase 1 Single Center, Open-Label, Randomized Two-Period, Two-Arm Crossover Study of the Relative Bioavailability of a Single Dose of CTP-543 in Fasted and Fed Conditions in Healthy Volunteers
Brief Title: Food Effect Study of CTP-543 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CP543.1003
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Safety; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: CTP-543 with meal Period 2: CTP-543 without meal
  Interventions: Drug: CTP-543
- Sequence 2 (Experimental): Period 1: CTP-543 without meal Period 2: CTP-543 with meal
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Once daily dosing

SUMMARY:
Two period crossover study to assess the bioavailability of CTP-543 under fed and fasted conditions.

DETAILED DESCRIPTION:
This open-label, single-dose study will assess in healthy subjects a solid oral dose formulation of CTP-543 under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 55 years of age, inclusive
* Body weight not less than 100 lbs and body mass index within the range of 18 to 32 kg/m2, inclusive, at screening

Exclusion Criteria:

* History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions
* PR interval > 220 msec or QRS duration > 120 msec or QTcF interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening
* Urinalysis positive for greater than trace blood, protein or glucose
* History of drug or alcohol abuse within 6 months of screening
* History of tobacco product use within 3 months prior to the study
* Inability to comply with dietary restrictions during study participation
* Blood donation or collection within 8 week prior to dosing
* Positive pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Measurement of CTP-543 in plasma under fed and fasted conditions | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States